CLINICAL TRIAL: NCT01307423
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) in Subjects With Active Psoriatic Arthritis Who Have Not Been Previously Treated With Disease-modifying Antirheumatic Drugs
Brief Title: Efficacy and Safety Study of Apremilast to Treat Active Psoriatic Arthritis (PsA)
Acronym: PALACE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-005; 2010-020324-22 (EudraCT Number)
Record Dates: First submitted 2010-11-29; First posted 2011-03-02 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: psoriasis; Arthritis; Psoriatic Arthritis; inflammation; skin condition; inflammatory cells; apremilast; CC-10004; phosphodiesterase type 4
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Arthritis; Inflammation; Skin Diseases | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Apremilast 20mg (Experimental): Apremilast 20mg twice daily, orally
  Interventions: Drug: Apremilast 20mg
- Apremilast 30mg (Experimental): Apremilast 30mg twice daily, orally
  Interventions: Drug: Apremilast 30mg
- Placebo + 20mg Apremilast (Placebo Comparator): Placebo + 20mg Apremilast tablets administered twice daily
  Interventions: Drug: Apremilast 20mg; Drug: Placebo
- Placebo + 30mg Apremilast (Placebo Comparator): Placebo + 30mg Apremilast tablets administered twice daily
  Interventions: Drug: Apremilast 30mg; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast 20mg — Apremilast 20mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 20mg; Placebo + 20mg Apremilast
Drug: Apremilast 30mg — Apremilast 30mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 30mg; Placebo + 30mg Apremilast
Drug: Placebo — Placebo
  Arms: Placebo + 20mg Apremilast; Placebo + 30mg Apremilast

SUMMARY:
The purpose of this study is to determine whether apremilast is safe and effective in the treatment of patients with psoriatic arthritis who have not been previously treated with DMARDs.

Apremilast is proposed to improve signs and symptoms of psoriatic arthritis (tender and swollen joints, pain, physical function) in treated patients.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is an inflammatory arthritis that occurs in 6-39% of psoriasis patients. The immunopathogenesis of PsA, which mirrors but is not identical to that seen in psoriatic plaques, reflects a complex interaction among resident dendritic, fibroblastic and endothelial cells, and inflammatory cells attracted to the synovium by cytokines and chemokines. Apremilast (CC-10004) is a novel oral agent that modulates multiple inflammatory pathways through targeted phosphodiesterase type 4 (PDE4) enzyme inhibition. Therefore, apremilast has the potential to be effective in the treatment of PsA.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Male or female, aged ≥ 18 years at time of consent.
2. Must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Have a documented diagnosis of Psoriatic Arthritis (PsA, by any criteria) of ≥ 3 months duration.
5. Meet the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria for PsA at time of screening.
6. Have ≥ 3 swollen AND ≥ 3 tender joints.
7. Have not been previously treated with disease-modifying antirheumatic drugs (DMARDS) (small molecules or biologics)
8. Be receiving treatment on an outpatient basis.
9. If taking oral corticosteroids, must be on a stable dose of prednisone ≤ 10 mg/day or equivalent for at least 1 month prior to screening.
10. If taking nonsteroidal anti-inflammatory drugs (NSAIDs) or narcotic analgesics, must be on stable dose for at least 2 weeks prior to screening and until they have completed the Week 24 study visit.
11. Low potency topical corticosteroids (Appendix M or locally available equivalent) will be allowed as background therapy for treatment of psoriasis on the face, axillae and groin in accordance with the manufacturers' suggested usage during the course of the study. Subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions. A non-medicated skin emollient (eg, Eucerin cream) will also be permitted for body lesions only. Subjects must not use these treatments within 24 hours prior to the clinic visit.
12. Meet the following laboratory criteria:

    * White blood cell count ≥ 3000/mm3 (≥ 3.0 x 109/L) and < 14,000/mm3 (< 14 x 109/L)
    * Platelet count ≥ 100,000/mm3 (≥ 100 x 109/L)
    * Serum creatinine ≤ 1.5 mg/dL(≤ 132.6 μmol/L)
    * Aspartate aminotransferase/Serum glutamic oxaloacetic transaminase (AST/SGOT) and Alanine aminotransferase/Serum glutamic pyruvic transaminase (ALT/SGPT) ≤ 2 x upper limit of normal (ULN)
    * Total bilirubin ≤ 2 mg/dL (≤ 34 μmol/L)
    * Hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L)
    * Hemoglobin A1c ≤ 9.0%
13. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex condom or any nonlatex condom NOT made out of natural [animal] membrane [eg, polyurethane]) while on IP and for at least 28 days after the last dose of IP.
14. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use 2 forms of contraception while on investigational product (IP) and for at least 28 days after the last dose of IP: one highly effective form (ie, hormonal, intrauterine device [IUD], tubal ligation, vasectomized partner) and one additional form (latex condom or any nonlatex condom NOT made out of natural [animal] membrane [eg, polyurethane], diaphragm, sponge). If one highly effective form of contraception cannot be used, then 2 forms of barrier contraception must be used, ie, latex condom or any nonlatex condom NOT made out of natural (animal) membrane (eg, polyurethane) with either of the following: sponge with spermicide or diaphragm with spermicide.

Exclusion Criteria:

1. History of clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease.
2. Any condition, including the presence of laboratory abnormalities that places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Clinically significant abnormality on 12-lead electrocardiography (ECG) at Screening.
4. Pregnant or breast feeding.
5. History of allergy to any component of the IP.
6. Hepatitis B surface antigen positive at screening.
7. Hepatitis C antibody positive at screening.
8. AST/SGOT and/or ALT/SGPT > 1.5 x ULN and total bilirubin > ULN or albumin < lower limit of normal (LLN).
9. History of positive Human Immunodeficiency Virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency Disease).
10. Active tuberculosis or a history of incompletely treated tuberculosis.
11. Clinically significant abnormality based upon chest radiograph with at least PA view (radiograph must be taken within 12 weeks prior to Screening or during the Screening visit). An additional lateral view is strongly recommended but not required.
12. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
13. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed at least 4 weeks prior to Screening.
14. Malignancy or history of malignancy (except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and treated [ie, cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix).
15. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
16. Erythrodermic, guttate, or pustular psoriasis.
17. Topical therapy for psoriasis, except as noted in the Inclusion Criteria, within 2 weeks of randomization (including but not limited to topical corticosteroids, topical retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin).
18. Rheumatic autoimmune disease other than PsA, including systemic lupus erythematosis (SLE), mixed connective tissue disease (MCTD), scleroderma, or polymyositis.
19. Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis (Appendix Q).
20. Prior history of or current inflammatory joint disease other than PsA (eg, gout, reactive arthritis, RA, ankylosing spondylitis, Lyme disease).
21. Prior use of disease modifying antirheumatic drugs (DMARDS; small molecules or biologics).
22. Use of the following systemic therapy(ies) within 4 weeks of randomization, including but not limited to corticosteroids (except as noted in inclusion criteria), oral retinoids and fumaric acid esters.
23. Use of phototherapy within 4 weeks of randomization (ie, UVB, PUVA).
24. Previous treatment with any cell depleting therapies, including investigational agents (eg, rituximab, CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19, and anti-CD20).
25. Treatment with intravenous gamma globulin, plasmapheresis, or Prosorba® column within 6 months of baseline.
26. Any previous treatment with alkylating agents such as cyclophosphamide or chlorambucil, or with total lymphoid irradiation.
27. Prior treatment with apremilast.
28. Use of any investigational drug within 4 weeks of randomization, or 5 pharmacokinetic/ pharmacodynamic half lives, if known (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2010-12-09 (Actual); Primary Completion 2013-02-21 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (118):
- United States (30):
  - Arizona Research Center, Phoenix, Arizona
  - Desert Medical Advances, Palm Desert, California
  - In Vivo Clinical Research, Doral, Florida
  - Centre For Rheumatology, Immun. And Arthritis, Fort Lauderdale, Florida
  - North Florida Dermatology, Jacksonville, Florida
  - Florida Center for Dermatology, PA, Saint Augustine, Florida
  - Tampa Medical Group Pa, Tampa, Florida
  - Atlanta Dermatology, Vein and Research Center, PC, Alpharetta, Georgia
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Sonora Clinical Research, LLC, Boise, Idaho
  - Rockford Orthopedic Associates, LLC, Rockford, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Indiana. University, Indianapolis, Indiana
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Justus Fiechtner MD PC, Lansing, Michigan
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Physicians East, Greenville, North Carolina
  - Unifour Medical Research Associatets LLC, Hickory, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Center for Clinical Studies, Houston, Texas
  - Houston Medical Research, Houston, Texas
  - Luckster Enterprises, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
  - PharmaSeek, Middleton, Wisconsin
- Australia (6):
  - Monash Medical Centre, Clayton, Victoria
  - Eastern Health Clinical School, Box Hill
  - Repatriation General Hospital, Daws Park
  - Menzies Centre for Population Health Research, Hobart
  - Optimus Clinical Research Pty. Ltd, Kogarah
  - The Queen Elizabeth Hospital, Woodville
- Belgium (2):
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Trimontsium, Plovdiv
  - 17 Diagnostic and Consulting Centre Sofia EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski, Sofia
  - Diagnostic-Consultative Center Sveta Anna, Sofia
  - Diagnostic Consulting Center N4, Varna
- Canada (12):
  - Arthritis Research Centre of Canada, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - St. Clare's Health Care Corporation of St. John's, St. John's, Newfoundland and Labrador
  - Ultranova Skincare, Barrie, Ontario
  - William Bensen's Private Practice, Hamilton, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Wilderman Medical Clinic, Thornhill, Ontario
  - Probity Medical Research Inc, Waterloo, Ontario
  - Darryl Toth's Private Practice, Windsor, Ontario
  - Centre de Rhumatologie St-Louis, Sainte-Foy, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- Czechia (4):
  - Revmatologicky ustav, Prague
  - Revmatologicka Ambulance, Prague
  - Affidea Praha s.r.o, Prague
  - PV - MEDICAL, s.r.o., Zlín
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Regional Hospital, Tallinn
  - Clinical Research Centre Ltd, Tartu
- France (4):
  - Hotel Dieu, Nantes
  - Groupe Hospitalier Archet I et II, Nice
  - Fondation Hôpital Saint-Joseph, Paris
  - Hopital Lariboisiere, Paris
- Hungary (7):
  - Qualiclinic kft, Budapest
  - Synexus Magyarország Kft., Budapest
  - Honvéd Kórház - Állami Egészségügyi Központ, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Principal SMO Kft., Makó
  - MAV Korhaz es Rendelointezet Szolnok, Szolnok
- Italy (5):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Ospedale Luigi Sacco, Milan
  - AOU della II Universita degli Studi di Napoli, Napoli
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Ospedale Civile Maggiore Borgo Trento, Verona
- Siauliai Hospital, Šiauliai, Lithuania
- New Zealand (3):
  - Waikato hospital, Hamilton
  - North Shore Hospital, Takapuna
  - Timaru Hospital, Timaru
- Poland (10):
  - Bytomskie Centrum Medyczne Silesiana Sp. z o.o., Bialystok
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Silesiana Sp. z o.o., Bytom
  - Synexus SCM Sp. z o.o., Gdynia
  - Synexus SCM Sp. z o.o., Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej REUMED, Lublin
  - Prywatna Praktyka Lekarska, Poznan
  - REUMATIKA-Centrum Reumatologii Niepubliczny Zaklad Opieki Zdrowotnej, Warsaw
  - Synexus SCM Sp. z o.o. Oddz. Warszawa, Warsaw
  - Synexus SCM Sp. z o.o., Wroclaw
- Romania (4):
  - Sf. Maria Clinical Hospital, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Sf Apostol Andrei Emergency Clinical County Hospital, Galati
  - C.M.I. Dr. Ciornohuz Adriana, Iași
- Russia (12):
  - Veterans of Wars Regional Clinical Hospital, Kemerovo
  - Kemerovo State Medical Academy of Roszdrav, Kemerovo
  - Research Medical Complex Vashe Zdorovie, Kezch
  - Krasnoyarsk State Medical Academy, Krasnoyarsk
  - City Clinical Hospital #5, Nizhny Novgorod
  - Research Institute of Clinical Immunology, Novosibirsk
  - Research Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - Departmental Hospital at Smolensk Station RZhD JSC, Smolensk
  - Tomsk Regional Clinical Hospital, Tomsk
  - Regional Clinical Hospital, Vladimir
  - Voronezh Regional Clinical Hopsital #1, Voronezh State Medical Academy, Voronezh
- South Korea (3):
  - Chungnam National University Hospital, Daejeon
  - Inha University Hosiptal, Incheon
  - Gachon University Gil Medical Center, Incheon
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Tapei
- United Kingdom (5):
  - Barnsley Hospital, Barnsley South Yorkshire
  - Haywood Hospital, Burslem
  - Cannock Chase Hospital, Cannock
  - Poole Hospital, Poole
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Mease PJ, Kavanaugh A, Ogdie A, Wells AF, Bergman M, Gladman DD, Richter S, Teng L, Jardon S, Smolen JS. Baseline Disease Activity Predicts Achievement of cDAPSA Treatment Targets With Apremilast: Phase III Results in DMARD-naive Patients With Psoriatic Arthritis. J Rheumatol. 2022 Jul;49(7):694-699. doi: 10.3899/jrheum.210906. Epub 2022 Apr 15. PMID 35428720
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Wells AF, Edwards CJ, Kivitz AJ, Bird P, Guerette B, Delev N, Paris M, Teng L, Aelion JA. Apremilast monotherapy for long-term treatment of active psoriatic arthritis in DMARD-naive patients. Rheumatology (Oxford). 2022 Mar 2;61(3):1035-1043. doi: 10.1093/rheumatology/keab449. PMID 34100922
- [Derived] Wells AF, Edwards CJ, Kivitz AJ, Bird P, Nguyen D, Paris M, Teng L, Aelion JA. Apremilast monotherapy in DMARD-naive psoriatic arthritis patients: results of the randomized, placebo-controlled PALACE 4 trial. Rheumatology (Oxford). 2018 Jul 1;57(7):1253-1263. doi: 10.1093/rheumatology/key032. PMID 29635379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 16 countries including the United States, Canada, Europe, New Zealand, Australia and Russia.
Pre-assignment Details: This study consisted of a 24-week randomized, double-blind, placebo-controlled phase, a 28-week randomized, double-blind active treatment phase and a 4-year open-label safety phase, for an overall study duration of 5 years.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily (BID) in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase and continued to receive 20 mg apremilast tablets twice daily for up to 4.5 years in the active treatment / long-term safety phase.
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase and continued to receive 30 mg apremilast tablets twice daily for up to 4.5 years in the active treatment / long-term safety phase.
- Placebo/ Apremilast 20 mg EE: Participants initially randomized to receive placebo twice daily who were re-randomized due to early escape (EE) at Week 16 to receive 20 mg apremilast twice daily in the active treatment phase.
- Placebo / Apremilast 20 mg XO: Participants initially randomized to receive placebo twice daily who were re-randomized at Week 24 (XO) to receive 20 mg apremilast twice daily in the active treatment phase.
- Placebo / Apremilast 30 mg EE: Participants initially randomized to receive placebo twice daily who were re-randomized due to early escape (EE) at Week 16 to receive 30 mg apremilast twice daily in the active treatment phase.
- Placebo / Apremilast 30 mg XO: Participants initially randomized to receive placebo twice daily who were re-randomized at Week 24 to receive 30 mg apremilast twice daily in the active treatment phase.
- Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)]: Participants initially randomized to placebo tablets twice daily during the 24-week placebo-controlled phase were re-randomized to 20 mg apremilast tablets twice daily at Week 16 or Week 24 and continued receiving apremilast 20 mg tablets twice daily in active treatment / long-term safety phase. (After 30 mg apremilast BID was identified as the optimal dose, all participants receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose).
- Placebo/Apremilast 30 mg (Long-Term Safety Phase): Participants initially randomized to placebo tablets BID during the 24-week placebo-controlled phase were re-randomized to apremilast 30 mg tablets twice daily at Week 16 or Week 24 and continued receiving apremilast 30 mg tablets twice daily in the active treatment / long-term safety phase.
Period: Placebo-controlled Phase (Week 0 - 24)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 176 | 175 | 177 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 176 | 175 | 175 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 166 | 168 | 166 | 0 | 0 | 0 | 0 | 0 | 0
Early Escape at Week 16 | 103 (One participant who escaped early did not complete Week 24) | 73 | 79 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 156 (Two participants did not escape early and finished Week 24 did not enter the active treatment phase) | 160 | 155 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 15 | 22 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization Error | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase (Week 25-52)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 151 (Nine participants who completed Week 24 did not enter active treatment phase) | 150 (Five participants who completed Week 24 did not enter active treatment phase) | 46 (Four participants who escaped early and completed Week 24 did not enter the active treatment phase.) | 26 | 46 (Six participants who escaped early and completed Week 24 did not enter the active treatment phase) | 26 | 0 | 0
Completed | 0 | 132 | 141 | 38 | 23 | 43 | 25 | 0 | 0
Not Completed | 0 | 19 | 9 | 8 | 3 | 3 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 5 | 5 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 11 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Long-term Safety Phase (Year 2)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 122 (10 participants who completed Week 52 did not enter the long-term safety phase) | 134 (7 participants who completed Week 52 did not enter the long-term safety phase) | 0 | 0 | 0 | 0 | 57 (Patients from the PBO/APR 20 mg EE and XO are combined;15 patients finished Wk 52;no entry into LTSP) | 67 (Patients from the PBO/APR 30 mg EE and XO are combined;5 patients finished Wk 52;no entry into LTSP)
Completed | 0 | 99 | 109 | 0 | 0 | 0 | 0 | 48 | 60
Not Completed | 0 | 23 | 25 | 0 | 0 | 0 | 0 | 9 | 7
Not completed — Adverse Event | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 7 | 5 | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Noncompliance with study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 13 | 12 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Miscellaneous | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Period: Long-term Safety Phase (Year 3)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started (The PBO/APR 20 mg and 30 mg EE and XO patients from week 24-52 are combined within the LTSP) | 0 | 99 | 109 | 0 | 0 | 0 | 0 | 48 | 60
Completed | 0 | 90 | 91 | 0 | 0 | 0 | 0 | 40 | 49
Not Completed | 0 | 9 | 18 | 0 | 0 | 0 | 0 | 8 | 11
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Lack of Efficacy | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Noncompliance with Study Drug | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 8 | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Miscellaneous | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Long-term Safety Phase (Year 4)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started (The PBO/APR 20 mg and 30 mg EE and XO patients from week 24-52 are combined within the LTSP) | 0 | 89 (1 participant who completed Year 3 did not continue treatment in Year 4) | 91 | 0 | 0 | 0 | 0 | 40 | 49
Completed | 0 | 81 | 86 | 0 | 0 | 0 | 0 | 38 | 44
Not Completed | 0 | 8 | 5 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 4 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Long-term Safety Phase (Year 5)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo/ Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg [Long-Term Safety Phase (LTSP)] | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started (The PBO/APR 20 mg and 30 mg EE and XO patients from week 24-52 are combined within the LTSP) | 0 | 81 | 86 | 0 | 0 | 0 | 0 | 38 | 44
Completed | 0 | 71 | 80 | 0 | 0 | 0 | 0 | 37 | 41
Not Completed | 0 | 10 | 6 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set was defined as participants who were randomized as specified in the protocol; one participant who was randomized in error and did not receive any dose of investigational product was excluded.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
- Apremilast 30mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg | Total
Number analyzed (Participants) | 176 | 175 | 176 | 527
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.58) | 49.2 (12.00) | 48.4 (12.52) | 49.4 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 95 | 96 | 277
  Male | 90 | 80 | 80 | 250
Duration of Psoriatic Arthritis [Mean (Standard Deviation); unit: years] — Psoriatic arthritis (PsA) is a chronic and progressive inflammatory arthritis that, depending on the method of ascertainment, occurs in 6% to 39% of patients with psoriasis. Disease onset typically occurs between the ages of 30 and 55 years and affects both sexes equally. In the majority of patients, psoriasis precedes PsA by several years. The diagnosis of PsA is made on clinical grounds in patients with psoriasis having skin, scalp or nail changes.
  years | 3.42 (5.103) | 3.19 (4.706) | 3.62 (5.041) | 3.41 (4.947)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: -Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); -Patient's global assessment of disease activity (measured on a 100 mm VAS); -Physician's global assessment of disease activity (measured on a 100 mm VAS); -Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); -C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: Full analysis set consisting of all participants randomized as specified in the protocol; one participant randomized in error and not receiving any dose of investigational product was excluded. Participants who withdrew early or did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 15.9 | 28.0 | 30.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; In order to maintain the Type 1 error at the 0.05 significance level, the Hochberg procedure was to be used. The results of the endpoint were to be considered statistically significant if both the 30 mg apremilast dose versus placebo comparison and the 20 mg versus placebo comparison were statistically significant at the 0.05 significance level, or one of the comparisons was statistically significant at the 0.025 level; Test type: Superiority or Other; p = 0.0062, Chi-squared; Risk Difference (RD) = 12.1, 95% CI 2-sided [3.5 to 20.7] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0010, Chi-squared; Risk Difference (RD) = 14.8, 95% CI 2-sided [6.1 to 23.5] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index [HAQ-DI]) at Week 16
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative changes from baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | 0.012 (0.0350) | -0.156 (0.0349) | -0.205 (0.0350)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Pairwise comparisons (30 mg vs placebo and 20 mg vs placebo) were conducted conditional on the primary endpoint results. If the primary endpoint was statistically significant for both apremilast dose groups, pairwise comparisons for the HAQ-DI were to be evaluated at the 0.05 level using the Hochberg procedure. If only one apremilast dose was statistically significant, then only the comparison between that apremilast dose and placebo was conducted for the HAQ-DI score, at the 0.025 level; Test type: Superiority or Other; p = 0.0008, ANCOVA; Based on an analysis of covariance (ANCOVA) model with treatment group as a factor, and the baseline value as a covariate; LS Mean Difference = -0.168, 95% CI 2-sided [-0.265 to -0.071]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.217, 95% CI 2-sided [-0.314 to -0.120]

3. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 13.1 | 29.1 | 24.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0002, Chi-squared — Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; Risk Difference (RD) = 16.1, 95% CI 2-sided [7.7 to 24.4] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0063, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 11.4, 95% CI 2-sided [3.3 to 19.4] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index [HAQ-DI]) at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Apremilast 20 mg: Participants initially randomized to receive Apremilast 20 mg tablets twice daily.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | 0.012 (0.0370) | -0.156 (0.0368) | -0.207 (0.0369)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0014, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Based on an analysis of covariance model for the change from baseline at Week 24, with treatment group as a factor and baseline value as a covariate; LS Mean Difference = -0.168, 95% CI 2-sided [-0.271 to -0.065]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.219, 95% CI 2-sided [-0.322 to -0.117]

5. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 16
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). SF-36 domain scores were first calculated to range from 0 to100 and then transformed to norm-based scores (the norm-based scores in the US general population have an average of 50 and a standard deviation of 10). Norm-based scores were used in analyses, with higher scores indicating a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | 0.01 (0.588) | 2.39 (0.586) | 3.19 (0.590)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0043, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Based on an analysis of covariance model for the change from baseline at Week 16, with treatment group as a factor and baseline value as a covariate; LS Mean Difference = 2.38, 95% CI 2-sided [0.75 to 4.01]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 3.18, 95% CI 2-sided [1.55 to 4.82]

6. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 16
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0=lowest disease activity and 100=highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0=lowest disease activity and 100=highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 16
Population: Full analysis set; Participants who discontinued early, or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 24.4 | 38.9 | 45.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0037, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 14.4, 95% CI 2-sided [4.8 to 24.0] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p < .0001, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 21.0, 95% CI 2-sided [11.3 to 30.7] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

7. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 16
Description: The participant was asked to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
mm | -2.6 (1.81) | -7.7 (1.79) | -10.5 (1.80)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0485, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -5.0, 95% CI 2-sided [-10.0 to -0.0]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0022, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -7.8, 95% CI 2-sided [-12.8 to -2.8]

8. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 115 | 117 | 111
units on a scale | -0.5 (0.24) | -0.5 (0.24) | -1.5 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.7696, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.6] — Based on an analysis of covariance model for the change from baseline at Week 16, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.7 to -0.3] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 16
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet will be rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline to Week 16
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 90 | 89 | 84
units on a scale | -1.0 (0.25) | -1.9 (0.25) | -1.7 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.9, 95% CI 2-sided [-1.6 to -0.2] — Based on analysis of covariance model for the change from baseline at Week 16, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.7, 95% CI 2-sided [-1.4 to -0.0] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 16
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 166 | 164
units on a scale | -1.98 (0.770) | -6.89 (0.763) | -7.63 (0.768)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -4.91, 95% CI 2-sided [-7.04 to -2.78] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -5.65, 95% CI 2-sided [-7.78 to -3.51] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) After 16 Weeks of Treatment
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 164 | 167
units on a scale | -0.15 (0.076) | -0.61 (0.076) | -0.68 (0.075)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.67 to -0.25] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.74 to -0.32] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 16
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 167 | 168 | 166
units on a scale | 0.07 (0.631) | 1.19 (0.629) | 2.62 (.0633)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Difference in LS Means = 1.12, 95% CI 2-sided [-0.63 to 2.87] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Difference in LS Means = 2.55, 95% CI 2-sided [0.80 to 4.31] — [estimate comment as in outcome 8, analysis 1]

13. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 24
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | 0.16 (0.609) | 2.13 (0.605) | 3.88 (0.611)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Means Difference = 1.97, 95% CI 2-sided [0.28 to 3.65] — Based on an analysis of covariance model for the change from baseline at Week 24, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 3.72, 95% CI 2-sided [2.02 to 5.41] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 24
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16, or who did not have sufficient data for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 20 mg: Participants initially randomized to receive Apremilast 20 mg tablets twice daily in the 24-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 17.0 | 36.6 | 35.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 19.5, 95% CI 2-sided [10.5 to 28.6] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 18.2, 95% CI 2-sided [9.2 to 27.2] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

15. Secondary Outcome: Change From Baseline in Participants Assessment of Pain at Week 24
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
mm | -3.8 (1.83) | -9.4 (1.82) | -9.6 (1.83)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -5.6, 95% CI 2-sided [-10.6 to -0.5] — Based on an analysis of covariance (Ancova) model for the change from baseline at Week 24, with treatment group as a factor and the baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -5.7, 95% CI 2-sided [-10.8 to -0.7] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 24
Description: as for outcome 8
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 111 | 113 | 106
units on a scale | -0.6 (0.25) | -0.9 (0.25) | -1.5 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.9, 95% CI 2-sided [-1.6 to -0.2] — [estimate comment as in outcome 15, analysis 1]

17. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 24 are included. LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 87 | 85 | 79
units on a scale | -1.0 (0.26) | -2.0 (0.26) | -1.7 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -1.0, 95% CI 2-sided [-1.7 to -0.3] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.6, 95% CI 2-sided [-1.4 to 0.1] — [estimate comment as in outcome 15, analysis 1]

18. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | -2.23 (0.807) | -7.30 (0.803) | -7.36 (0.810)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -5.07, 95% CI 2-sided [-7.31 to -2.84] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -5.14, 95% CI 2-sided [-7.38 to -2.89] — Based on an analysis of covariance model (Ancova) for the change from baseline at Week 24, with treatment group as a factor and the baseline value as a covariate

19. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS 28) at Week 24
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | -0.22 (0.084) | -0.69 (0.084) | -0.68 (0.084)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.70 to -0.23] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.69 to -0.22] — [estimate comment as in outcome 18, analysis 2]

20. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
units on a scale | 0.25 (0.652) | 1.37 (0.648) | 2.58 (0.655)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 1.12, 95% CI 2-sided [-0.68 to 2.93] — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean difference = 2.33, 95% CI 2-sided [0.52 to 4.15] — [estimate comment as in outcome 18, analysis 2]

21. Secondary Outcome: Percentage of Participants With ≥ 20% Improvement in Maastricht Ankylosing Spondylitis Entheses Score at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 115 | 117 | 111
percentage of participants | 46.1 | 48.7 | 63.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.6, 95% CI 2-sided [-10.2 to 15.5] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 17.0, 95% CI 2-sided [4.2 to 29.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

22. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 90 | 89 | 84
percentage of participants | 60.0 | 66.3 | 61.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.3, 95% CI 2-sided [-7.8 to 20.4] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 1.9, 95% CI 2-sided [-12.6 to 16.4] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

23. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Week 16
Description: The EULAR response criteria classify each subject as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease. Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 25.0 | 41.1 | 44.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 16.1, 95% CI 2-sided [6.4 to 25.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 19.3, 95% CI 2-sided [9.6 to 29.1] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

24. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 115 | 117 | 111
percentage of participants | 48.7 | 54.7 | 66.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.0, 95% CI 2-sided [-6.8 to 18.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 18.0, 95% CI 2-sided [5.3 to 30.6] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

25. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 90 | 89 | 84
percentage of participants | 57.8 | 69.7 | 63.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 11.9, 95% CI 2-sided [-2.1 to 25.9] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 5.3, 95% CI 2-sided [-9.2 to 19.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

26. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response at Week 24
Description: The EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on th DAS-28. Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2 A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 17.0 | 34.9 | 28.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 17.8, 95% CI 2-sided [8.8 to 26.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 11.4, 95% CI 2-sided [2.7 to 20.0] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

27. Secondary Outcome: Percentage of Participants With a ACR 50 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Groups:
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
Percentage of participants | 4.5 | 11.4 | 11.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.9, 95% CI 2-sided [1.3 to 12.5] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.8, 95% CI 2-sided [1.2 to 12.4] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

28. Secondary Outcome: Percentage of Participants With a ACR 70 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 1.1 | 4.0 | 4.0
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.9, 95% CI 2-sided [-0.4 to 6.2] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.8, 95% CI 2-sided [-0.4 to 6.1] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

29. Secondary Outcome: Percentage of Participants With a ACR 50 Response at Week 24
Description: as for outcome 27
Time Frame: Baseline and Week 24
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 6.3 | 16.0 | 12.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 9.8, 95% CI 2-sided [3.2 to 16.3] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.3, 95% CI 2-sided [0.2 to 12.3] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

30. Secondary Outcome: Percentage of Participants With a ACR 70 Response at Week 24
Description: as for outcome 28
Time Frame: Baseline and Week 24
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30mg
Number analyzed (Participants) | 176 | 175 | 176
percentage of participants | 4.0 | 4.0 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 0.0, 95% CI 2-sided [-4.1 to 4.1] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; Risk Difference (RD) = 0.6, 95% CI 2-sided [-3.7 to 4.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

31. Secondary Outcome: Percentage of Participants With Pre-existing Enthesopathy Whose Maastricht Ankylosing Spondylitis Entheses Score Improves to 0 at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 115 | 117 | 111
percentage of participants | 19.1 | 21.4 | 36.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 2.2, 95% CI 2-sided [-8.1 to 12.6] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 17.8, 95% CI 2-sided [6.3 to 29.3] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

32. Secondary Outcome: Percentage of Participants With Pre-existing Dactylitis Whose Dactylitis Severity Score Improves to 0 at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30mg
Number analyzed (Participants) | 90 | 89 | 84
percentage of participants | 33.3 | 42.7 | 40.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 9.4, 95% CI 2-sided [-4.8 to 23.5] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; Risk Difference (RD) = 7.1, 95% CI 2-sided [-7.2 to 21.5] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

33. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 24
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 115 | 117 | 111
percentage of participants | 22.6 | 29.1 | 37.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Risk Difference (RD) = 6.5, 95% CI 2-sided [-4.8 to 17.7] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.4 to 27.1] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

34. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 90 | 89 | 84
percentage of participants | 35.6 | 46.1 | 40.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 10.5, 95% CI 2-sided [-3.8 to 24.8] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Risk Difference (RD) = 4.9, 95% CI 2-sided [-9.5 to 19.3] — Two-sided 95% CI of the proportion difference is based on the normal approximation to the binomial distribution

35. Secondary Outcome: Percentage of Participants With a ACR 20 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: ≥ 20% improvement in 78 tender joint count; ≥ 20% improvement in 76 swollen joint count; and ≥ 20% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population consists of all participants who were randomized or re-randomized to apremilast at any time during the study. Only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Placebo / Apremilast 20 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 20 mg apremilast twice daily.
- Placebo / Apremilast 30 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 30 mg apremilast twice daily.
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily.
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 67 | 131 | 138
Percentage of Participants | 59.7 [46.4 to 71.9] | 56.7 [44.0 to 68.8] | 53.4 [44.5 to 62.2] | 58.7 [50.0 to 67.0]

36. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 68 | 132 | 139
units on a scale | -0.21 (0.450) | -0.25 (0.533) | -0.32 (0.559) | -0.39 (0.567)

37. Secondary Outcome: Change From Baseline in the SF-36v2 Physical Functioning Scale Score at Week 52
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 68 | 132 | 139
units on a scale | 7.76 (8.236) | 6.87 (7.241) | 5.68 (8.467) | 5.87 (8.008)

38. Secondary Outcome: Percentage of Participants With a Modified PsARC Response at Week 52
Description: Measure Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0=lowest disease activity and 100=highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0=lowest disease activity and 100=highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 61 | 67 | 131 | 139
Percentage of Participants | 73.8 [60.9 to 84.2] | 79.1 [67.4 to 88.1] | 75.6 [67.3 to 82.7] | 75.9 [67.9 to 82.8]

39. Secondary Outcome: Change From Baseline in the Participants Assessment of Pain Using the Visual Analog Scale at Week 52
Description: as for outcome 7
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo/Apremilast 20 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 20 mg apremilast twice daily.
Arm/Group | Placebo/Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 68 | 132 | 139
mm | -13.1 (25.57) | -18.9 (24.28) | -15.6 (27.29) | -14.2 (28.14)

40. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 52
Description: as for outcome 8
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo/Apremilast 30 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 30 mg apremilast twice daily.
Arm/Group | Placebo / Apremilast 20 mg | Placebo/Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 41 | 42 | 91 | 176
units on a scale | -1.7 (2.38) | -1.8 (2.34) | -1.5 (2.62) | -1.8 (3.03)

41. Secondary Outcome: Change From Baseline in the Dactylitis Severity Score at Week 52
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing dactylitis) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 32 | 38 | 70 | 64
units on a scale | -2.2 (1.89) | -2.9 (2.47) | -2.2 (4.09) | -2.9 (3.55)

42. Secondary Outcome: Change From Baseline in the CDAI Score at Week 52
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: 28 tender joint count (TJC), 28 swollen joint count (SJC), Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 61 | 67 | 131 | 137
units on a scale | -11.0 (10.288) | -14.67 (11.943) | -14.32 (11.128) | -13.98 (10.541)

43. Secondary Outcome: Change From Baseline in the DAS28 at Week 52
Description: as for outcome 11
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 68 | 130 | 138
units on a scale | -1.08 (1.113) | -1.28 (1.044) | -1.37 (1.128) | -1.39 (0.970)

44. Secondary Outcome: Change From Baseline in the FACIT-Fatigue Scale Score at Week 52
Description: as for outcome 12
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 67 | 131 | 139
units on a scale | 6.03 (8.787) | 4.27 (9.461) | 2.39 (10.197) | 5.89 (10.471)

45. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 52 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 41 | 42 | 91 | 85
Percentage of Participants | 70.7 [54.5 to 83.9] | 81.0 [65.9 to 91.4] | 65.9 [55.3 to 75.5] | 69.4 [58.5 to 79.0]

46. Secondary Outcome: Percentage of Participants With Pre-existing Dactylitis Whose Dactylitis Severity Score Improves From Baseline by ≥ 1 at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 32 | 38 | 70 | 64
Percentage of Participants | 93.8 [79.2 to 99.2] | 94.7 [82.3 to 99.4] | 87.1 [77.0 to 93.9] | 85.9 [75.0 to 93.4]

47. Secondary Outcome: Percentage of Participants Achieving Good or Moderate EULAR Response at Week 52
Description: The EULAR response criteria classify each subject as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease. A Good response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 A Moderate Response is defined as either: an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2. Two-sided 95% confidence interval is based on the Clopper-Pearson method
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 68 | 130 | 138
Percentage of Participants | 64.5 | 73.5 | 75.4 | 79.0

48. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: ≥ 50% improvement in 78 tender joint count; ≥ 50% improvement in 76 swollen joint count; and ≥ 50% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 67 | 129 | 138
Percentage of Participants | 30.6 [19.6 to 43.7] | 25.4 [15.5 to 37.5] | 27.1 [19.7 to 35.7] | 31.9 [24.2 to 40.4]

49. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 52
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: ≥ 70% improvement in 78 tender joint count; ≥ 70% improvement in 76 swollen joint count; and ≥ 70% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 61 | 68 | 131 | 138
Percentage of Participants | 8.2 [2.7 to 18.1] | 10.3 [4.2 to 20.1] | 13.7 [8.4 to 20.8] | 18.1 [12.1 to 25.6]

50. Secondary Outcome: Percentage of Participants With Pre-existing Enthesopathy Whose MASES Improves From Baseline to 0 at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Achilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval was based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 41 | 42 | 91 | 85
percentage of participants | 39.0 [24.2 to 55.5] | 61.9 [45.6 to 76.4] | 39.6 [29.5 to 50.4] | 45.9 [35.0 to 57.0]

51. Secondary Outcome: Percentage of Participants With Pre-existing Dactylitis Whose Dactylitis Severity Score Improves From Baseline to 0 at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit and ranges from 0 to 20. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 46
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 32 | 38 | 70 | 64
Percentage of Participants | 75.0 [56.6 to 88.5] | 78.9 [62.7 to 90.4] | 68.6 [56.4 to 79.1] | 68.8 [55.9 to 79.8]

52. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Placebo Controlled Phase
Description: A TEAE is an adverse event (AE) with a start date on or after the date of the first dose of investigational product (IP) and no later than 28 days after the last dose of IP. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. A serious AE is any AE that results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or constitutes an important medical event. For both AEs and SAEs the investigator assessed the severity of the event according to the grading scale: Mild: asymptomatic or with mild symptoms, Moderate: symptoms causing moderate discomfort or Severe: symptoms causing severe discomfort or pain.
Time Frame: Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants (placebo participants who remained on placebo through week 24 and participants randomized to the APR 20 mg BID or APR 30 mg BID)
Population: Safety population included participants who were randomized and received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 176 | 175 | 175
Participants
  Any TEAE | 73 | 87 | 99
  Any Drug-Related TEAE | 25 | 40 | 58
  Any Severe TEAE | 6 | 4 | 2
  Any Serious TEAE (SAE) | 5 | 3 | 1
  Drug-Related (SAE) | 0 | 0 | 1
  Any TEAE Leading to Drug Interruption | 8 | 11 | 9
  Any TEAE Leading to Drug Withdrawal | 4 | 4 | 6
  Any TEAE Leading to Death | 0 | 0 | 0

53. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Apremilast Exposure Period
Description: as for outcome 52
Time Frame: Week 0 to Week 260; median duration of exposure to apremilast 20 mg BID was 168.93 weeks and 229.36 weeks for apremilast 30 mg BID
Population: Apremilast Subjects as Treated (AAT) were those who received at least 1 dose of apremilast at any time during the study. Participants were included in the treatment group corresponding to the apremilast dosing regimen they actually received, irrespective of the treatment group to which they were randomized or re-randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast 20 mg (Pre-Switch): Participants who received 20 mg apremilast tablets twice daily, regardless of when the apremilast exposure started (at Week 0, 16 or 24). Only the TEAEs that occurred during apremilast 20 mg BID were counted.
- Apremilast 20/30 mg (Post-Switch): Participants who switched from apremilast 20 mg tablets twice daily to apremilast 30 mg twice daily. Only the TEAEs that occurred during the apremilast 30 mg treatment were included.
- Apremilast 30 mg: Participants who received apremilast 30 mg twice daily regardless of when the apremilast-exposure started (at Week 0, 16, or 24).
Arm/Group | Apremilast 20 mg (Pre-Switch) | Apremilast 20/30 mg (Post-Switch) | Apremilast 30 mg
Number analyzed (Participants) | 252 | 122 | 252
Participants
  Any TEAE | 188 | 60 | 204
  Any Drug-Related TEAE | 89 | 16 | 113
  Any Severe TEAE | 24 | 3 | 23
  Any Serious TEAE (SAE) | 35 | 5 | 36
  Drug-Related (SAE) | 6 | 1 | 6
  Any TEAE Leading to Drug Interruption | 41 | 5 | 36
  Any TEAE Leading to Drug Wirhdrawal | 22 | 2 | 26
  Any TEAE Leading to Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs are reported for the placebo-controlled phase from Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants and reported for the Apremilast Exposure Period from Week 0 to Week 260; median duration of apremilast 20 mg BID was 168.93 weeks and 229.36 weeks for apremilast 30 mg twice daily
Groups:
- Weeks 0-24: Placebo (Placebo-Controlled Phase): Participants received placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 16 for participants who escaped early, and through Week 24 for all other participants.
- Weeks 0-24: Apremilast 20 mg: Participants received 20 mg apremilast tablets PO twice daily during the 24-week placebo-controlled phase.
- Weeks 0-24: Apremilast 30 mg: Participants received 30 mg apremilast tablets PO twice daily during the 24-week placebo-controlled phase.
- APR Exposure Period Up to 5 Years: Apremilast 20 mg: Participants who received apremilast 20 mg twice daily regardless of when the apremilast exposure started (at Week 0, 16 or 24). Only TEAEs that occurred during apremilast 20 mg BID treatment (before the switch to 30 mg apremilast) were included.
- APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg: Participants who switched from apremilast 20 mg twice daily to apremilast 30 mg BID. Only the TEAEs that occurred during apremilast 30 mg twice daily treatment were included.
- APR Exposure Period Up to 5 Years: Apremilast 30 mg: Participants who received apremilast 30 mg twice daily throughout the study regardless of when the apremilast exposure started (at Week 0, 16, or 24).
Arm/Group | Weeks 0-24: Placebo (Placebo-Controlled Phase) | Weeks 0-24: Apremilast 20 mg | Weeks 0-24: Apremilast 30 mg | APR Exposure Period Up to 5 Years: Apremilast 20 mg | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg | APR Exposure Period Up to 5 Years: Apremilast 30 mg
Serious Adverse Events (participants affected / at risk) | 5/176 | 3/175 | 1/175 | 35/252 | 5/122 | 36/252
Other Adverse Events (participants affected / at risk) | 30/176 | 51/175 | 65/175 | 121/252 | 24/122 | 141/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=176) | Weeks 0-24: Apremilast 20 mg (N=175) | Weeks 0-24: Apremilast 30 mg (N=175) | APR Exposure Period Up to 5 Years: Apremilast 20 mg (N=252) | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg (N=122) | APR Exposure Period Up to 5 Years: Apremilast 30 mg (N=252)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocele (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
Vertigo CNS origin (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Endometrial atrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=176) | Weeks 0-24: Apremilast 20 mg (N=175) | Weeks 0-24: Apremilast 30 mg (N=175) | APR Exposure Period Up to 5 Years: Apremilast 20 mg (N=252) | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg (N=122) | APR Exposure Period Up to 5 Years: Apremilast 30 mg (N=252)
Diarrhoea (Gastrointestinal disorders) | 3 | 12 | 21 | 30 | 2 | 31
Dyspepsia (Gastrointestinal disorders) | 2 | 8 | 0 | 14 | 0 | 4
Nausea (Gastrointestinal disorders) | 5 | 16 | 28 | 24 | 2 | 39
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 20 | 5 | 23
Sinusitis (Infections and infestations) | 1 | 6 | 4 | 16 | 6 | 12
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 7 | 26 | 5 | 31
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 10 | 3 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 14 | 0 | 10
Headache (Nervous system disorders) | 4 | 6 | 15 | 15 | 0 | 26
Depression (Psychiatric disorders) | 1 | 1 | 2 | 5 | 2 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 4 | 11 | 1 | 13
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 6 | 1 | 13
Hypertension (Vascular disorders) | 1 | 4 | 4 | 15 | 0 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.